CLINICAL TRIAL: NCT00001456
Title: Clinical and Basic Investigations Into Hermansky-Pudlak Syndrome
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950193; 95-HG-0193
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01-08

CONDITIONS: Hermansky-Pudlak Syndrome (HPS)
Keywords: Albinism; Platelet Storage Pool Deficiency; Metabolic Disease; Pulmonary Fibrosis; Inflammatory Bowel Disease; Natural History
MeSH Terms: conditions — Hermanski-Pudlak Syndrome; Albinism; Platelet Storage Pool Deficiency; Metabolic Diseases; Pulmonary Fibrosis; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HPS: HPS patients of any sex and ethnicity age 1-80 years
- HPS Symptom Questionnaire: Includes both patients and family members or caregivers.

SUMMARY:
Hermansky-Pudlak Syndrome (HPS) is an inherited disease which results in decreased pigmentation (oculocutaneous albinism), bleeding problems due to a platelet abnormality (platelet storage pool defect), and storage of an abnormal fat-protein compound (lysosomal accumulation of ceroid lipofuscin).

The disease can cause poor functioning of the lungs, intestine, kidneys, or heart. The major complication of the disease is pulmonary fibrosis and typically causes death in patients ages 40 - 50 years old. The disorder is common in Puerto Rico, where many of the clinical research studies on the disease have been conducted. Neither the full extent of the disease nor the basic cause of the disease is known. There is no known treatment for HPS.

The purpose of this study is to perform research into the medical complications of HPS and begin to understand what causes these complications. Researchers will clinically evaluate patients with HPS of all ethnic backgrounds. They will obtain cells, blood components (plasma), and urine for future studies. Genetic tests (mutation analysis) to detect HPS-causing genes will also be conducted.<TAB>...

DETAILED DESCRIPTION:
Study Description:

Hermansky-Pudlak syndrome is a rare autosomal recessive disease consisting of oculocutaneous albinism, a platelet storage pool defect and, in some patients, lysosomal accumulation of ceroid lipofuscin. Other manifestations include pulmonary fibrosis (often fatal in the fourth or fifth decade), chronic granulomatous colitis and, rarely, renal involvement or cardiomyopathy. The purpose of this protocol is to evaluate individuals with HPS, perform mutation analysis for known HPS-causing genes, search for variants in other genes responsible for HPS, and obtain specimens to analyze basic mechanisms of HPS.

Objectives:

Primary Objective: Assess the clinical severity of HPS, to study the natural history of disease, to identify variants in genes associated with HPS, and to investigate basic defect(s) in HPS and mechanisms of disease.

Study Population:

All participants will be persons with HPS, or their family members, aged 1-80 years. The enrollment ceiling is 600; we estimate that approximately 200 subjects will participate only in the HPS Symptom Questionnaire. Family members who are caregivers of affected individuals, including children, may be invited to participate in the HPS Symptom Questionnaire to provide responses related to their affected relative. We anticipate enrolling 2-10 new subjects per year under this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA

Persons with HPS or family members who are their caregivers aged 1-80 years are eligible to enroll in this protocol. The diagnosis of HPS is based upon a paucity or deficiency of platelet dense bodies on whole mount electron microscopy or the identification of pathogenic variants in HPS genes by genetic testing. Some persons who have not been diagnosed with HPS may be admitted to the protocol based upon the presence of albinism and a platelet storage pool deficiency.

Subjects participating only in the HPS Symptom Questionnaire will be at least 18 years of age.

EXCLUSION CRITERIA

Pregnant women and adults who are unable to provide consent are excluded.

Ages: 1 Month to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HPS patients of any sex and ethnicity age 1-80 years
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 1995-11-06 (Actual)

PRIMARY OUTCOMES:
Natural History | Ongoing
  The natural history of Hermansky-Pudlak Syndrome (HPS)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Introne, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
pending

REFERENCES:
- [Derived] Han CG, O'Brien KJ, Coon LM, Majerus JA, Huryn LA, Haroutunian SG, Moka N, Introne WJ, Macnamara E, Gahl WA, Malicdan MCV, Chen D, Krishnan K, Gochuico BR. Severe bleeding with subclinical oculocutaneous albinism in a patient with a novel HPS6 missense variant. Am J Med Genet A. 2018 Dec;176(12):2819-2823. doi: 10.1002/ajmg.a.40514. Epub 2018 Oct 4. PMID 30369044
- [Derived] El-Chemaly S, Cheung F, Kotliarov Y, O'Brien KJ, Gahl WA, Chen J, Perl SY, Biancotto A, Gochuico BR. The Immunome in Two Inherited Forms of Pulmonary Fibrosis. Front Immunol. 2018 Jan 31;9:76. doi: 10.3389/fimmu.2018.00076. eCollection 2018. PMID 29445374
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1995-HG-0193.html